CLINICAL TRIAL: NCT05992714
Title: The Effect of Virtual Rain Forest and White Noise on Satisfaction, Tolerance, Comfort and Vital Signs During Arthroscopy
Brief Title: Effects of VR and White Noise During Arthroscopy (VR/WN_ ART)
Acronym: (VR/WN_ ART)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seher Tanrıverdi (Other)
Responsible Party: Sponsor-Investigator, Seher Tanrıverdi, Asistant Professor, Mardin Artuklu University
Organization: Mardin Artuklu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: vr/white noise
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Arthroscopic Surgical Procedures
Keywords: virtual reality; tolerance; satisfaction; comfort; white noise
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Parallel Assignment experimental model using randomized pretest and posttest with control group
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Glasses (Experimental): Except for the preparation of the patient for the procedure, since the arthroscopy procedure takes approximately 60 minutes, 60-minute 360-degree VR video scenes will be watched using VR head device
  Interventions: Device: Virtual Reality Glasses group
- White Noise (Experimental): Except for the preparation of the patient for the procedure, since the arthroscopy procedure takes approximately 60 minutes, 60-minute 360-degree VR video scenes will be listened using phone
  Interventions: Device: white noise group
- control group (No Intervention): Patients of the control group, will not receive any intervention except for applied routine hospital arthroscopy surgery procedures

INTERVENTIONS:
Device: Virtual Reality Glasses group — Except for the preparation of the patient for the procedure, since the arthroscopy procedure takes approximately 60 minutes, 60-minute 360-degree VR video scenes will be watched using VR head device
  Arms: Virtual Reality Glasses
Device: white noise group — Except for the preparation of the patient for the procedure, since the arthroscopy procedure takes approximately 60 minutes, 60-minute 360-degree VR video scenes will be watched using phone
  Arms: White Noise

SUMMARY:
Background: Today, arthroscopy is widely used in the diagnosis and of treatment intra-articular diseases. Arthroscopy is considered a procedure that disturbs the patient's comfort because it is a very invasive and painful procedure especially spinal anesthesia. Along with physical discomfort during the procedure, it triggers, fear and anxiety in the patient.

Purpose: To examine the effects of virtual rain forest and white noise on patient satisfaction, pain, comfort and vital signs in patients of arthroscopic knee surgery.

Method: The population of the study consisted of all patients who applied to the Dicle University Hospital Orthopedics and Traumatology unit and were scheduled for arthroscopy in the operating room. Based on the sample size of Basak and Sahin's study using similar VR applications, 31 patients were determined for each group total 93 patients with 5% significance level and 80% power(13). G*Power, version 3.0.10 was used for statistical power analysis. The study group of 93 people to participate in the study will be divided into three equal groups in accordance with the random numbers table obtained the computer- based Research Randomizer program. Before the arthroscopy procedure, the patients included in the study will be randomly divided into three groups: 31 rain forest video VR group, 31 white noise group and 31 control group. Data will be collected in the in the operating room on weekdays when the procedure is performed.

ELIGIBILITY:
Inclusion Criteria:

18 aged and over, Written and verbal consent to participate in the study, Being conscious (person, place and time orientation), Undergoing colonoscopy for the first time Spinal anesthesia applied, Meniscus surgery will be performed patients.

Exclusion Criteria:

Having vision, hearing and communication problems, Having any psychiatric and cognitive/mental mental health problems, disease (dementia, etc.), Diagnosed with visual, auditory and / or balance disorders, General anesthesia applied patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Patient Information Form | the fundamental characteristics of the patients will be filled in 10 minutes before the arthroscopy procedure
  This form, which was created by the researcher; patients' age, gender, education level, marital status, employment status, income level, ASA level, chronic disease status, and previous surgery. It consists of a total of 9 questions
Visual Analogue Scale (VAS) | Change from Baseline Visual Analogue Scale in 1 hour
  This scale developed by Price (1983) will be used in the research to determine the level of tolerance, comfort and satisfaction. It is a scale in which the distance between the two ends with a minimum value of 0 on one end and a maximum value of 10 on the other end is measured with a 10 cm ruler. In this context; The patient is explained that there are two endpoints and that he is free to mark any place between them that fits the severity of his pain.
  The distance between the beginning of "no comfort, tolerance and satisfaction" and this point marked by the patient is measured and recorded in centimeters. It has been shown that the VAS is a valid tool for the measurement of psychological and health variables such as pain and satisfaction, which is widely used in clinical studies.
The Patient Observation Form | Change from Baseline The Patient Observation Form in 1 hour
  This form, which was created by the researcher, the vital signs (pulse, respiratory rate, systolic blood pressure (SBP), diastolic blood pressure (DBP), and oxygen saturation values (SpO2) of the patients before and after the procedure were recorded the form.

IPD SHARING:
Plan to Share IPD: Undecided
Undecided all IPD that underlie results in a publication

REFERENCES:
- [Background] Sahin G, Basak T. The Effects of Intraoperative Progressive Muscle Relaxation and Virtual Reality Application on Anxiety, Vital Signs, and Satisfaction: A Randomized Controlled Trial. J Perianesth Nurs. 2020 Jun;35(3):269-276. doi: 10.1016/j.jopan.2019.11.002. Epub 2020 Mar 4. PMID 32146074
- [Background] Celebi D, Yilmaz E, Sahin ST, Baydur H. The effect of music therapy during colonoscopy on pain, anxiety and patient comfort: A randomized controlled trial. Complement Ther Clin Pract. 2020 Feb;38:101084. doi: 10.1016/j.ctcp.2019.101084. Epub 2019 Dec 23. PMID 32056820
- [Background] Huang MY, Scharf S, Chan PY. Effects of immersive virtual reality therapy on intravenous patient-controlled sedation during orthopaedic surgery under regional anesthesia: A randomized controlled trial. PLoS One. 2020 Feb 24;15(2):e0229320. doi: 10.1371/journal.pone.0229320. eCollection 2020. PMID 32092098
- [Background] Umezawa S, Higurashi T, Uchiyama S, Sakai E, Ohkubo H, Endo H, Nonaka T, Nakajima A. Visual distraction alone for the improvement of colonoscopy-related pain and satisfaction. World J Gastroenterol. 2015 Apr 21;21(15):4707-14. doi: 10.3748/wjg.v21.i15.4707. PMID 25914482
- [Background] Veldhuijzen G, Klaassen NJM, Van Wezel RJA, Drenth JPH, Van Esch AA. Virtual reality distraction for patients to relieve pain and discomfort during colonoscopy. Endosc Int Open. 2020 Jul;8(7):E959-E966. doi: 10.1055/a-1178-9289. Epub 2020 Jun 30. PMID 32626819
- [Background] Ilkkaya NK, Ustun FE, Sener EB, Kaya C, Ustun YB, Koksal E, Kocamanoglu IS, Ozkan F. The effects of music, white noise, and ambient noise on sedation and anxiety in patients under spinal anesthesia during surgery. J Perianesth Nurs. 2014 Oct;29(5):418-26. doi: 10.1016/j.jopan.2014.05.008. PMID 25261145
- [Derived] Genc H, Tanriverdi S, Sait Akar M. The effect of virtual rainforest and a white noise mobile application on satisfaction, tolerance, comfort, and vital signs during arthroscopy. Complement Ther Clin Pract. 2024 May;55:101848. doi: 10.1016/j.ctcp.2024.101848. Epub 2024 Mar 15. PMID 38507879